CLINICAL TRIAL: NCT04532879
Title: HygiRelief Procedure and HygiSample Evaluation for Patients Diagnosed With Rome IV Functional Constipation Previously Managed With Linzess
Brief Title: HygiRelief Procedure and HygiSample Evaluation for Functional Constipation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: decided not to do the study due to Covid staffing restrictions
Sponsor: HyGIeaCare, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGP-0009
Record Dates: First submitted 2020-08-20; First posted 2020-08-31 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Rome IV Functional Constipation

STUDY DESIGN:
Intervention Model Description: Prospective, single center, open label. Patients will serve as their own control by comparing their bowel habits using a specific diary 2 weeks after the Linzess washout period to the 2 weeks after their HygiRelief procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- All patients enrolled (Experimental): Bowel habits before and after the HygiRelief procedure will be assessed.
  Samples will be sent for microbiome evaluation.
  Interventions: Device: HygiPrep (HyGIeaCare System)

INTERVENTIONS:
Device: HygiPrep (HyGIeaCare System) — Controlled gravity-based high-volume colon irrigation
  Other Names: HygiSample (stool collection for microbiome evaluation)

SUMMARY:
This study has a single center, prospective, open label design. The population will include patients diagnosed with Rome IV Functional Constipation who are at the time of study enrollment being managed with a stable dose of Linzess. They will stop taking their Linzess, undergo monitoring of bowel habits for 2 weeks, have a HygiRelief procedure and then undergo an additional 2 weeks of bowel habit monitoring.

DETAILED DESCRIPTION:
After undergoing a 5-7 day Linzess washout period, patients will record their bowel habits in a daily diary for 2 weeks. Patients will have the HygiRelief procedure with a HygiSample evaluation, then they will record their bowel habits in a daily diary for 2 weeks following the HygiRelief procedure.

HygiSamples (stool samples) will be collected throughout the HygiRelief procedure and the samples will be sent for microbiome evaluation.

Patients will complete multiple questionnaires - Happiness Scale, Hospital Anxiety and Depression Scale (HADS), and a personal assessment which includes the Constipation Symptom Score and Adverse Event Screening. These will be completed at Baseline, after the 2 week PRE-HygiRelief period, and after the 2 week POST-HygiRelief period.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age is between 18 and 80 years old
2. Patient diagnosed with Rome IV Functional Constipation (Attachment C2)
3. Patient is currently managed with Linzess and willing to stop taking it for study duration

Exclusion Criteria:

1. Patient has functional bowel disorders characterized by alternating bowel habits (diarrhea/constipation)
2. Patient has any other condition that, in the opinion of the investigator, may adversely affect the compliance or safety of the patient or would limit the patient's ability to complete the study
3. Patient has any of the contraindications listed below:

   1. Cardiac: Congestive heart failure (NYHA class III or IV or EF <50%)
   2. GI: Intestinal perforation, carcinoma of the rectum, fissures or fistula, severe hemorrhoids, abdominal hernia, recent colon, rectal, or abdominal surgery
   3. GU: Renal insufficiency (CC < 60 ml/min/173m2), cirrhosis with ascites
   4. Abdominal surgery within the last 6 months
   5. Pregnancy
4. Patient took antibiotics within two months of starting the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Assess change in bowel movements PRE and POST HygiRelief procedure | 12 months
  Evaluate the clinical effectiveness of the HygiRelief procedure to relieve functional constipation in patients previously managed with a stable dose of Lizess

SECONDARY OUTCOMES:
Assess colon effluent samples (HygiSample) collected during the HygiRelief procedure | 12 months
  Samples will be evaluated for their microbiological and biochemical content, as well as to identify microbiome changes throughout the colon

IPD SHARING:
Plan to Share IPD: No